CLINICAL TRIAL: NCT05848388
Title: Prevelance of Molar Incisor Malformation in Egypt
Brief Title: Molar Incisor Malformation in Egypt
Status: Completed | Type: Observational
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Maha Moussa Azab, Lecturer, Fayoum University
Other Study IDs: Molar Incisor Malformation
Record Dates: First submitted 2023-04-28; First posted 2023-05-08 (Actual); Last update posted 2023-05-08 (Actual); Status verified 2023-04

CONDITIONS: Paediatric Dentistry
Keywords: molar-incisor malformation, developmental malformation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: older than 9-year-old patients, with panoramic radiographic images showing the first permanent molars
  Interventions: Other: Molar incisor malformation presence

INTERVENTIONS:
Other: Molar incisor malformation presence — the presence of radiographic features of molar incisor malformation

SUMMARY:
The aim of the current study is to assess the prevalence of molar incisor malformation in Fayoum-Egypt.

DETAILED DESCRIPTION:
Localized developmental radicular dysplasia is a rare finding. This radicular formation arrest may be due to traumas, infections, radiation therapy, chemotherapy, or idiopathic.

Molar Incisor Malformation is a condition characterized by arrested or altered radicular development of first permanent molars. Roots may be thin, short, or totally missing. In some patients, there are constrictions located in the cervical part of the crown of the permanent incisors. There are also cases where the roots of the second primary molars are affected.

MIM could also have been mistaken for a consequence of severe root resorption, or dentine dysplasia prior to its initial description.

This unique deformity, regardless of its nomenclature, presents previously undescribed clinical features and it is quite difficult to get a successful conservative treatment result.

The aim of the current study is to assess the prevalence of this rare condition in Fayoum-Egypt.

ELIGIBILITY:
Inclusion Criteria:

* Panoramic radiographs for older than nine-year-old patients, having completely developed first permanent molars

Exclusion Criteria:

* Panoramic radiographs with missing first permanent molars or pathological lesions which may cause root resorption

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: panoramic radiographic images from a private dental radiology center in Fayoum Egypt
Sampling Method: Non-Probability Sample
Enrollment: 5630 (Actual)
Dates: Start 2022-05-30 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
molar incisor malformation | Day 1
  the presence of root malformation to indicate the diagnosis of molar incisor malformation

CONTACTS AND LOCATIONS:
Overall Officials: maha M azab, Principal Investigator — Fayoum University
Locations (1):
- Alpha Dent, Al Fayyum, Egypt